CLINICAL TRIAL: NCT01654835
Title: A Effectiveness Trial of Early Hemodynamic Support in Patients Demonstrating a Low Systolic Blood Pressure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 12-587
Record Dates: First submitted 2012-07-17; First posted 2012-08-01 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Intraoperative Low Blood Pressure
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low blood pressure alert (Active Comparator): A Low Blood Pressure condition as specified (SAP <80 mmHg)will trigger an page to be sent to all anesthesia providers in <1 min that will read: "A Low Blood Pressure condition has been detected. Consider hemodynamic support."
  Interventions: Other: low blood pressure alert
- no low blood pressure alert (Placebo Comparator): The Low Blood Pressure condition will be monitored by treatment team, but additional alert will not be sent to treatment team.
  Interventions: Other: standard of care

INTERVENTIONS:
Other: low blood pressure alert — A Low Blood Pressure condition as specified (SAP <80 mmHg)will trigger an page to be sent to all anesthesia providers in <1 min that will read: "A Low Blood Pressure condition has been detected. Consider hemodynamic support."
  Arms: low blood pressure alert
Other: standard of care — A Low Blood Pressure condition as specified (SAP <80 mmHg)will be monitored by treatment team upon detection, but additional paged alert will not be generated.
  Arms: no low blood pressure alert

SUMMARY:
The investigators thus propose to use an innovative randomized effectiveness trial design to test the theory that early automatic identification of a ¡ Low Systolic Blood Pressure¡± clinical condition and decision-support alerts will prompt earlier hemodynamic support and a consequently reduce the duration of such conditions. Specifically, the investigators will test the hypothesis that providing DSS alerts in regards to hypotension reduces the duration of hypotensive episodes. The core of the investigators study will be an existing electronic anesthesia record and smart-alarm decision-support system. All patients undergoing surgery at Hillcrest will be randomly assigned to routine care or to DSS support. In patients assigned to DSS support, a systolic blood pressure less than 80 mmHg will generate a warning within three minutes after detection. Clinicians will be free to act on the alert, ignore the alert, or to consider the provided information without acting on it. The randomization, complete anesthesia record, detailed record of hypotensive events, alerts provided, clinician responses, and SAP response, will be captured by the investigators electronic record-keeping system. The investigators primary outcome will be the duration of time the patient has a systolic blood pressure less than 80 mmHg. Secondary outcome will be duration of hospitalization. The investigators will assess the effect of the alert on the primary outcome of time to SBP returning to above 80 mmHg using survival analysis, with time to event censored (and considered a non-event) at either the end of surgery or end of monitoring if patient did not return to above 80 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be enrolled in the study if systolic blood pressure (SBP) is measured to be below 80 mmHg for at least 3 minutes, either with the arterial line or cuff (non-invasive blood pressure, NIBP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
duration of time having low blood pressure | day 1
  We plan to test the hypothesis that providing hypotension alerts reduces the duration of time patients spend in a low blood pressure condition.

SECONDARY OUTCOMES:
hypotension | day 1
  Secondary outcome will be the incidence of hypotension as well as duration of hospitalization
duration of hospitalization | up to day 3
  Secondary outcome will be the incidence of hypotension as well as duration of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Hillcrest Hospital Cleveland Clinic, Cleveland, Ohio, United States